CLINICAL TRIAL: NCT04992832
Title: Multi-intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells for Treatment in Heart Failure Patients With Reduced Ejection Fraction: A Randomized, Double Blind, Placebo-Controlled, Prospective Clinical Study
Brief Title: Multi-intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells in Heart Failure With Reduced Ejection Fraction（PRIME-HFrEF Study）
Acronym: PRIME-HFrEF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFSC-2018(CR)-08
Record Dates: First submitted 2021-07-13; First posted 2021-08-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure, Systolic
Keywords: Human Umbilical Cord Mesenchymal Stem Cells; Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The volunteers of the experimental group will be given peripheral intravenously a dose of 1.0*10^6/kg human umbilical cord mesenchymal stem cells at 0,6,12 week.
  Interventions: Biological: human umbilical cord mesenchymal stem cells
- control group (Placebo Comparator): The control group will be given the same dose of saline containing human albumin.
  Interventions: Other: human serum albumin

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — Human umbilical cord mesenchymal stem cells were peripheral intravenous infused to experimental group.
  Arms: experimental group
Other: human serum albumin — Saline solution containing 1 percent human serum albumin will be infused to the control group.
  Arms: control group

SUMMARY:
This study is an exploratory clinical study to observe the safety and efficacy of the Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells in the heart failure patients with reduced ejection fraction. The study was a 12 months single center, randomized, double-blind, placebo-controlled trial that included 12 weeks of treatment, and 9 months of follow-up.

DETAILED DESCRIPTION:
The study was a 12-month single center, randomized, double-blind, placebo-controlled trial that included 12 weeks of treatment, and 9 months of follow-up.We plan to recruit 40 subjects，which were divided into experimental group and control group. The volunteers of the experimental group will be given peripheral intravenously infusion a dose of 1.0*10^6/kg human umbilical cord mesenchymal stem cell (HUC-MSC) respectively at 0,6,12 week. The control group will be given the same dose of 1 percent human serum albumin injection. Then centralization visit was conducted at 0,7 day, 6,12 week, 6 and 12 month. The primary safety end point is the incidence of any treatment emergent serious adverse events within12 months after intravenous MSC infusion, including death, nonfatal MI, stroke, sustained ventricular arrhythmias (>15 seconds or causing hemodynamic compromise), and other adverse events such as infection, tumor formation and clinical abnormal, which will be evaluated by monitoring for serial troponin, hematology, chemistry, urinalysis, 24-hour Holter, CTscans and ultrasound of abdomen.There are independent data and safety monitoring committees to monitor patient safety throughout the duration the trial.The primary efficacy endpoint is a change in Left Ventricular Ejection Fractions (LVEF) measured by left ventricular opacification (LVO) with contrast echocardiography and magnetic resonance imaging (MRI) at 12th month.

ELIGIBILITY:
Inclusion Criteria:

1. LVEF≤40％;
2. NYHA II-IV;
3. Received maximally tolerated guideline-directed medical therapy ( GDMT) for at least 3 months before enrollment;
4. Angiography or coronary CT within 6 months shows that there is no indication for PCI / CABG; Or PCI / CABG indications, but refused.

Exclusion Criteria:

1. Severe valvular heart disease, congenital heart disease, acute viral myocarditis and acute coronary syndrome.
2. PCI / CABG, ICD / permanent pacemaker / CRT implantation within 3 months.
3. Recent cerebrovascular disease (<6 months).
4. eGFR<30ml/min, or ALT/AST>120U/L.
5. Hematologic disease: anemia (hemoglobin ≤9.0 g/dL); leukopenia (<3500/μL); thrombocytopenia (<70000/μL); myeloproliferative disorders, myelodysplastic syndrome, acute or chronic leukemia, and plasma cell dyscrasias (multiple myeloma, amyloidosis) .
6. Malignant tumor within 5 years.
7. Life expectancy <1 year according any disease.
8. Uncontrolled acute infectious diseases.
9. Known or suspected of being sensitive to the study drugs or its ingredients.
10. Not suitable for inclusion according to the evaluation of the sponsors or unwilling to comply with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
The safety of treatment | Day 360
  The incidence of treatment related adverse events
Left ventricular ejection fraction | Day 360
  The change in Left ventricular ejection fraction (LVEF) % after the infusion.

SECONDARY OUTCOMES:
A composite of cardiac death and rehospitalization caused by heart failure within 12 months | 12 month after treatment
  The comparison of the mortality and the incidence of rehospitalization caused by heart failure between the two groups.
NT-proBNP | Day 360
  The change in NT-proBNP after the infusion.
ST2 | Day 360
  The change in ST2 after the infusion.
Left ventricular end systolic volume | Day 43, Day 85, Day 180, Day 360
  The change in Left ventricular end systolic volume(LVESV) after the infusion
6 minutes walking distance | Day 360
  The change in 6 minutes walking distance after the infusion.
The SUV in PET-MR | Day 180
  The change of standard uptake value in PET-MR after the infusion
Right ventricular end systolic volume | Day 360
  The change in Right ventricular end systolic volume(RVESV) after the infusion
Tricuspid annular plane systolic excursion | Day 360
  Changes of Right ventricular tricuspid annular plane systolic excursion (TAPSE) detected by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Liu, Doctor, Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Heart Failure Department, East Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided